CLINICAL TRIAL: NCT05900778
Title: Implementation of a HABIT-ILE Intervention at William Lennox Neurological : a Randomized Controlled Trial
Brief Title: Implementation of a HABIT-ILE Intervention at William Lennox Neurological Hospital (NeuREHA)
Acronym: NeuREHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B0392023000044
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Acquired Brain Injury
Keywords: motor skill learning; executive function; activity of daily living; intensive therapy; acquired brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): Hand and arm bimanuel intensive therapy including lowers extremities
  Interventions: Behavioral: HABIT-ILE
- Conventional intervention (Active Comparator): Conventional physical and occupational therapy
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: HABIT-ILE — 2 weeks HABIT-ILE
  Arms: HABIT-ILE
Behavioral: Conventional intervention — 2 weeks usual intervention (waitlist group)
  Arms: Conventional intervention

SUMMARY:
Using a randomized controlled trial design, in an hospital environment, possible changes induced by the "Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)" treatment program will be investigated in functional activities of daily living, motor and cognitive assessment of children with acquired brain injury.

DETAILED DESCRIPTION:
The aim is to investigate, for the first time, the effectiveness of HABIT-ILE therapy in a hospital setting in the treatment of a population representative of the clinical population with children with acquired brain injuries.

The hypothesis is that an in-hospital HABIT-ILE protocol will be more effective than conventional therapies usually given to children with acquired brain injury, and that this difference will be objectively demonstrated by clinical assessments of motor function, cognition and participation conducted before and after treatment periods.

The aim of the study is therefore to evaluate the effect of intensive bimanual hand-arm therapy including the lower extremities (HABIT-ILE) on body functions and structures, activity and participation in children with acquired brain injury.

ELIGIBILITY:
Inclusion Criteria:

* children with acquired brain injury of school
* age 5 to 18 years inclusive

Exclusion Criteria:

* Unstable seizure
* programmed botulinum toxin or orthopedic surgery in the 6 months previous to the intervention, during intervention period or 3months after the intervention time
* Severe visual or cognitive impairments likely to interfere with intervention or testing session completion

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Flanker task | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  Cognitive functions of the children will be assessed by Flanker task.
Changes in Gross Motor Function Measurement (GMFM 66) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The GMFM has been developed to measure the change in gross motor function over time in children with cerebral palsy.

SECONDARY OUTCOMES:
Changes in isometric muscular strength (Jamar) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  A quantitative and objective measure of isometric muscular strength of hand and forearm.
Stroop task | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  Executive functions of the children will be assessed by Stroop task.
Changes in unimanual dexterity: Box and Blocks test (BBT) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The BBT is a test of gross manual dexterity. Each hand is tested individually and the BBT is scored through the number of blocks carried over the partition from one part to another part of a box during the one-minute trial period.
Changes on bimanual function (Assisting Hand Assessment (AHA)) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  Developed to observe the efficacy of the assisting hand use, in children with unilateral cerebral palsy (scored in percentage), during bimanual activities for the randomized controlled trial
Changes in 6 Minutes Walking Test (6MWT) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The 6 Minutes Walking Test measures the distance that the patient walk as much as possible within a period of 6-minutes in a 30 meters long corridor.
Changes in Pediatric balance scale (PBS) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  A 14-item criterion-referencekd measure that examines functional balance in the context of everyday tasks in the pediatric population.
Changes in Canadian Occupational Performance Measure (COPM) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  This is an interview-setting designed to capture a patient's self-perception of performance and satisfaction of it in everyday activities, observed over time. During the interview, parents set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the child's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10; higher score means better performance/satisfaction)
Changes in ACTIVLIM-CP questionnaire | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  This parent's filled questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower extremities through 43 items specific to patients with cerebral palsy. It ranges from - 7 to +7 logits (higher score means better performance).
Changes in Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The PEDI-CAT is the new version of the Pediatric Evaluation of Disability Inventory (PEDI). The PEDI-CAT is comprised of 276 functional activities acquired throughout infancy, childhood and young adulthood. Based on the nternational Classification of Functioning, Disability and Health for Children and Youth (ICF-CY) model, the PEDI-CAT contents provide information about the activities and participation component. It ranges from 0 to 100% (higher score means better performance).
Changes in Pediatric quality of life inventory (PedsQL) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The Pediatric Quality of Life Inventory is a brief measure of health-related quality of life in children and young people. The measure can be completed by parents (the Proxy Report) as well as children and young people (the Self-Report).
Changes in Measure of Processes of Care (MPOC-20) | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  Assesses the parents' perceptions of the care they and their children receive from children's rehabilitation treatment centres. Using a 8-point response scale, parents answer to 20 questions, indicating to what extent they have experienced the events or the situations described. A score of 7 means that they have experienced this aspect to a very great extent, or most of the time. A score of 1 means that they have not experienced this aspect at all. A score of 0 means that the question does not apply to them.
  There is no total score. However, because the statements are positively worded, higher total scores indicates that needs of the parents are being met to a great extent.
Status in Wechsler Intelligence Scale for Children-Non verbal short version (WISC) | T0 (baseline)
  This is a validated assessment for children aged 4 and over, with subtests such as object assembly, recognition, picture arrangement and fluid reasoning. The brief 15-20 minute version will be used. Scores are given for the full battery and for the subtests (subtest T-scores and percentile ranks).
Classification du niveau moteur: The Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R) | T0 (baseline)
  The Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R) is a 5-level classification system that describes the gross motor function of children and youth on the basis of their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility.
QUALITY OF LIFE : KIDSCREEN 10 | T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, Professor, Principal Investigator — Insititue of Neurosciences, UCLouvain
Locations (3):
- Belgium (3):
  - Centre Hospitalier Neurologique William Lennox, Ottignies-Louvain-la-Neuve, Brabant-Wallon
  - Institute of Neurosciences, UCLouvain, Brussels
  - Spontaneous contact via doctors or other partners, Brussels

IPD SHARING:
Plan to Share IPD: No